CLINICAL TRIAL: NCT06464913
Title: A Randomized Phase II Trial on Omission of Chest Wall Radiotherapy After Implant-Based Breast Reconstruction in Early Breast Cancer Patients
Brief Title: Randomized Phase II Trial: Chest Wall RT Omission After Prosthetic Reconstruction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y2024-0423
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms
Keywords: Post-mastectomy radiation therapy; Implant-based breast reconstruction; Local recurrence; Reconstruction failure
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: Open-label design, where the assessors are not blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Chest Wall RT (Experimental): This group will have chest wall RT omitted and will only receive RT to the supraclavicular and infraclavicular lymphatic drainage areas.
  Interventions: Radiation: With or without chest wall RT
- Traditional RT (Active Comparator): This group will receive standard RT to the chest wall and supraclavicular and infraclavicular lymphatic drainage areas.
  Interventions: Radiation: With or without chest wall RT

INTERVENTIONS:
Radiation: With or without chest wall RT — Supraclavicular and infraclavicular lymphatic drainage area radiotherapy with or without chest wall RT

SUMMARY:
The goal of this randomized Phase II clinical trial is to test the effects of omitting chest wall radiotherapy (RT) after prosthetic reconstruction in early-stage breast cancer patients. The main questions it aims to answer are:

* Can omitting chest wall RT after prosthetic reconstruction reduce the failure rate of breast reconstruction without significantly increasing the local recurrence rate?
* Does this approach ensure an improvement in the quality of life for patients without sacrificing therapeutic effectiveness?

Participants will:

* Be randomly assigned to one of two groups.
* One group will receive standard RT to the chest wall and supraclavicular and infraclavicular lymphatic drainage areas.
* The other group will have chest wall RT omitted and will only receive RT to the supraclavicular and infraclavicular lymphatic drainage areas.
* Participate in follow-up assessments to monitor reconstruction failure rates and local recurrence rates.

If there is a comparison group: Researchers will compare the outcomes of the two groups to evaluate the impact of chest wall RT omission on reconstruction failure and local recurrence risks.

DETAILED DESCRIPTION:
Breast reconstruction, as part of the surgical treatment for breast cancer, offers an opportunity for patients who have undergone mastectomy to restore their body image and mental state, while post-mastectomy radiation therapy (PMRT) has advantages in local control and long-term survival of breast cancer. However, the integration of PMRT with reconstruction, especially using implants, raises concerns due to potential complications and the risk of reconstruction failure.

Reconstruction methods include autologous tissue and prosthetic implants, with the latter becoming more popular due to shorter surgery times and faster recovery. The choice between immediate, delayed, and two-stage reconstruction depends on tumor characteristics and patient factors. PMRT indications are based on tumor features and risks. The 2019 ESTRO expert consensus pointed out that the radiotherapy target area after breast prosthetic implantation should include the chest wall and all high-risk lymphatic drainage areas of the axillary region that have not been removed. While PMRT improves outcomes, it increases complications in implant-based reconstructions. Within two years after prosthetic reconstruction surgery, the proportion of patients who have at least one complication after radiotherapy is 39%, while it is 22% for patients who have not received radiotherapy. Early complications include fat or flap necrosis, thrombosis, infection, hematoma, delayed wound healing, and late complications include pain, prosthetic contracture, prosthetic exposure or rupture, and a decline in various indicators of aesthetic results. Patients who ultimately have to remove the implant or convert to autologous tissue reconstruction due to severe complications are defined as reconstruction failure. Among patients who received implant reconstruction and radiotherapy, the proportion of reconstruction failure after two years is the highest (18.7%); in contrast, the failure rate in the non-radiotherapy group or autologous reconstruction group is less than 5%.

Considering the high incidence of complications after prosthetic implantation, the failure rate of breast reconstruction may exceed 20%, while the local recurrence rate after breast reconstruction surgery is around 5%. For early-stage breast cancer patients undergoing cold knife one-step prosthetic reconstruction or two-step expander-prosthetic reconstruction, whether omitting chest wall radiotherapy can reduce the failure of reconstruction without significantly increasing the local recurrence rate, to ensure that improving the quality of life for patients does not sacrifice therapeutic effects. In response to this issue, this project proposes a "randomized Phase II clinical trial of omitting chest wall radiotherapy after prosthetic reconstruction in early-stage breast cancer" prospective study. This study will adopt a randomized controlled method, dividing patients into two groups, one group receiving routine chest wall plus supraclavicular and infraclavicular lymphatic drainage area radiotherapy, and the other group omitting chest wall radiotherapy and only receiving supraclavicular and infraclavicular lymphatic drainage area radiotherapy, aiming to evaluate the impact of omitting chest wall radiotherapy in PMRT after prosthetic reconstruction on the reconstruction failure rate of breast cancer patients, without significantly increasing the risk of local recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Undergoes prosthetic reconstruction (including cold knife one-step prosthetic reconstruction or two-step expander-prosthetic reconstruction.);
* Histologically confirmed invasive breast cancer patients with stage T1-2N1M0;
* ECOG score of 0-1;
* Indications for neoadjuvant therapy before surgery and adjuvant therapy after surgery.

Exclusion Criteria:

* Other metabolically active malignant tumors;
* Severe dysfunction of heart, lung, liver, kidney, or other vital organs;
* Uncontrolled diabetes or other endocrine diseases;
* Known allergy to radiotherapy or chemotherapy drugs;
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Reconstruction failure rate (Capsular Contracture Grade III or higher) | 2 years postoperatively
  Physicians assess the hardness, shape of the breast, and the presence of any abnormal hard lumps or asymmetry through palpation. According to the Baker classification system, capsular contracture is divided into four grades; Grades I and II typically have no clinical significance, while Grades III and IV require further evaluation and possible treatment.
  Breast Ultrasound or Chest CT is used to assess the condition of the implant and surrounding tissues. Particularly, the thickening of the fibrous capsule is considered an objective sign of capsular contracture.
  In cases where the results of the ultrasound examination are unclear or a more detailed assessment is needed, MRI may be required to evaluate the implant and surrounding tissues.
The 3-year local recurrence rate (LRR) | 3 years postoperatively
  The 3-year LRR refers to the proportion of patients who experience a cancer recurrence within the breast tissue or chest wall area, or in the regional lymph nodes, within three years following the initial treatment.
  To determine the local recurrence rate, medical professionals:
  Conduct regular follow-up examinations, including physical assessments and patient-reported symptoms.
  Utilize imaging techniques such as mammography, ultrasound, computed tomography (CT), or magnetic resonance imaging (MRI) when indicated.
  May also consider the use of tumor markers in blood tests to monitor for signs of recurrence.

SECONDARY OUTCOMES:
Breast-Q score | 2 years postoperatively
  The Breast-Q score is a patient-reported outcome measure (PROM) specifically designed to assess the satisfaction and quality of life of patients who have undergone breast surgery.The questionnaire assesses multiple dimensions, including body image, pain, sexual life, and satisfaction, to comprehensively reflect the quality of life and the success of postoperative surgery for patients. Patients self-assess based on the questions in the scale, with each question usually having multiple levels to choose from, and different scores are assigned according to the level selected. The total score is obtained by summing the scores of all questions. The higher the Breast-Q score, the better the patient's quality of life and the greater the satisfaction with the surgery.
PROs and QoL score | 3 years postoperatively
  Satisfaction score (patient-reported outcome) and Quality of Life (QoL) score Measurement Method: A questionnaire is designed based on the assessment dimensions of the patient's physical function, mental health, social function, pain, satisfaction, body image, sexual function, etc., including multiple-choice questions, single-choice questions, scale scoring (such as VAS), open-ended questions, etc.
3-year disease free survival rate (DFS) | 3 years postoperatively
  The 3-year DFS rate refers to a percentage of patients who are disease-free at the three-year mark after their initial treatment. Researcher conduct regular follow-up assessments, including physical examinations and patient-reported outcomes. Utilize imaging studies such as mammograms, CT scans, MRI, or PET scans when appropriate. Monitor for any signs or symptoms that may indicate a recurrence of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No